CLINICAL TRIAL: NCT06876311
Title: Sponsor-initiated, Retrospective, Monocentric, Non-interventional Clinical Observational Study to Evaluate the STALIF® C FLX, STALIF® M FLX, STALIF® L FLX Cages and FORTOS-C®
Brief Title: Observational Study to Evaluate the STALIF® C FLX, STALIF® M FLX, STALIF® L FLX Cages and FORTOS-C®
Status: Active, not recruiting | Type: Observational
Sponsor: Silony Medical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TDI_2023_004_2.1_103
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Degenerative Cervical Disc Disease; Degenerative Lumbar Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- FORTOS-C: Patients treated with FORTOS-C
  Interventions: Device: Anterior Cervical Interbody Fusion
- STALIF C FLX: Patients treated with STALIF C FLX
  Interventions: Device: Anterior Cervical Interbody Fusion
- STALIF M FLX: Patients treated with STALIF M FLX
  Interventions: Device: Anterior lumbar Interbody Fusion
- STALIF L FLX: Patients treated with STALIF L FLX
  Interventions: Device: Lateral Lumbar Interbody Fusion

INTERVENTIONS:
Device: Anterior Cervical Interbody Fusion — Standard Anterior Cervical Interbody Fusion with Stand-alone Cervical Cages
  Groups: FORTOS-C; STALIF C FLX
Device: Anterior lumbar Interbody Fusion — Standard Anterior Lumbar Interbody Fusion with Stand-Alone Lumbar Cages
  Groups: STALIF M FLX
Device: Lateral Lumbar Interbody Fusion — Standard Lateral Lumbar Interbody Fusion with Stand-alone Lumbar cage
  Groups: STALIF L FLX

SUMMARY:
Post-operative clinical outcome data on the devices used to treat spinal diseases are collected and evaluated in order to analyze the safety and performance of the implants used.

ELIGIBILITY:
Inclusion Criteria:

- Indications according to IFU

Surgical implantation of STALIF® C or M FLX device for 1 or 2 levels between:

* STALIF® C FLX: C2-T1 (cervical)
* STALIF® M FLX: L2-S1 (lumbar)
* STALIF® L FLX: L2-L5 (lumbar)

Surgical implantation of FORTOS-C® for the fusion of up to 3 levels between:

* FORTOS-C®: C2 - T1 (cervical)
* Age: ≥ 21 years
* For the evaluation of the questionnaires (NDI or ODI, VAS neck and VAS arm or VAS leg and VAS back), only patients with the questionnaire available at the time of admission (pre-op) and at least at 12-months FU will be included

Exclusion Criteria:

* Relative and absolute contraindications according to IFU

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population is defined by Inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | Baseline, 3 months postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The Neck Disability Index (NDI) has 10 items that cover various aspects of daily functioning, such as pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
  Scoring: Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst. Alternately, the score can be reported from 0-100. The score is often reported as a percentage (0-100%).
Oswestry Disability Index | Baseline, 3 months postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The Oswestry Disability Index (ODI) is used to measure the extent of pain-related functional limitations in people with low back pain. The questionnaire provides the user with information about the general functional ability of a patient with low back pain in everyday life. Six response options are available for the following items: pain intensity, self-care (washing, dressing), lifting, locomotion, sitting or standing, sleeping, sex life, social life and travel/transportation. The first answer option (score 0) means that there are no pain-related restrictions, while the sixth answer option (score 5) indicates the greatest perceived restriction of an activity due to pain.

SECONDARY OUTCOMES:
Visual Analogue Scale | Baseline, 3 months postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The Visual Analogue Scale (VAS) is usually quantified from 0 to 10, where 0 means 'no pain' and 10 means 'strongest pain imaginable'.
Radiological assessment | Baseline, 3 months postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  * Implant migration/ Subsidence/ Screw Back-out
  * Bone Fusion at latest follow-up
Complications | Baseline, 3 months postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  Intraoperative and postoperative complications, revisions, and (serious) adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Golden State Orthopedics and Spine, San Ramon, California, United States

IPD SHARING:
Plan to Share IPD: No